CLINICAL TRIAL: NCT03266523
Title: Pilot Study on the Influence of the Integration of Natural Images, According to Various Esthetic Approaches, in the Waiting Rooms of Imaging on the Anxiety Felt by the Patients
Brief Title: Influence of Natural Images on Patients' Anxiety in the Waiting Rooms of Imaging Ward
Acronym: VERTIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/49
Record Dates: First submitted 2017-07-12; First posted 2017-08-30 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: All Conditions for Which a CT or MRI Exam Can be Required
Keywords: CT; MRI; Anxiety-state; Anxiety State-Trait
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: The CONTROL (neutral) environment corresponds to the standard environment of the imaging waiting rooms
- Zen: The ZEN environment will represent a clean, minimalist nature
  Interventions: Other: Natural images in imaging waiting rooms
- Green: The GREEN environment will represent rural landscapes, undergrowth
  Interventions: Other: Natural images in imaging waiting rooms
- Sea: The SEA environment will represent lakes, ponds, seaside
  Interventions: Other: Natural images in imaging waiting rooms

INTERVENTIONS:
Other: Natural images in imaging waiting rooms — Standard environment for hospital imaging waiting rooms
  Other Names: Neutral
  Groups: Green; Sea; Zen

SUMMARY:
VERTIM study aims to evaluate the influence of different environments of imaging waiting rooms on the anxiety felt by patients before MRI or CT scans. For this, four environments (neutral/standard; and nature "green", "sea", and "zen") will be set up in MRI and CT waiting rooms.

DETAILED DESCRIPTION:
Each year, the Medical Imaging Unit of the University Hospital of Bordeaux (CHU Bordeaux) receives 80,500 patients for CT or MRI scans in usual care. The length of waiting, the environment of the waiting room, the reasons for the examination are factors that increase the levels of anxiety during waiting and but also during early examination.

Previous studies have shown that the integration of nature (real as well as artificial) is likely to decrease the level of anxiety. Before implementing a multicentre and randomised trial, a pilot study is necessary to assess the feasibility of the procedure, to test the relevance of the tools, to identify the influence of socio-cultural and socio-demographic characteristics on anxiety's level.

For this, the present study will be conducted over the same period of the year in order to avoid seasonality biases. The study will take place over 8 weeks, during which MRI or scanner patients will be exposed either to the neutral environment (standard environment of the waiting room) or to one of the 3 environments (wall posters representing the nature ("green", "sea", "zen")).

There is no specific intervention assigned to the study participants, i.e. the patients will receive one of the four environments as part of routine medical care, and a researcher studies the effect of this environment on anxiety's level. Every week, one environment will be set up in the MRI or scanner waiting room and the study will be proposed to all eligible patients present in this room. Fifty patients are expected each week so that 100 patients per environment and equally distributed between the MRI and scanner waiting rooms are expected.

ELIGIBILITY:
Inclusion Criteria:

* patient 18 yrs and older;
* patients in MRI or scanner's waiting room awaiting one of these 2 exams;
* patients not objecting to answer questionnaires;
* patient covered under social security

Exclusion Criteria:

* patient <18yrs old;
* patients with hearing and visual impairments;
* patients unable to answer questionnaires;
* patients awaiting for other exams than MRI or scanner;
* legally protected patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are major patients who will be present in the waiting room of the MRI or the scanner in order to carry out one of these two exams
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Average of the scores of anxiety-State (STAI-Y). | The day the patient waits in the imaging waiting room

SECONDARY OUTCOMES:
Average of the scores of emotional perception for the various esthetic approaches | The day the patient waits in the imaging waiting room
Scores of the anxiety-trait in each of the subgroups | The day the patient waits in the imaging waiting room
Scores of satisfaction for the various esthetic approaches | The day the patient waits in the imaging waiting room
Strength of the interaction between emotional perception *environnement to explain the level of anxiety State | The day the patient waits in the imaging waiting room
  This outcome is measured through the scores of emotional perception (emotional perception), the nature of environment applied (control, zen, green or sea) and the STAI-Y scale score (level of state anxiety)
Reliability of the tool: coefficient alpha of Cronbach, or coefficient α ≥ 0,7. | The day the patient waits in the imaging waiting room
Reason for MRI or scanner's prescription | The day the patient waits in the imaging waiting room
Anxiolytic treatment and / or antidepressants (regular intake) | The day the patient waits in the imaging waiting room
Anxiolytic treatment (specific prescription for examination) | The day the patient waits in the imaging waiting room
gender | The day the patient waits in the imaging waiting room
age | The day the patient waits in the imaging waiting room
Level of education | The day the patient waits in the imaging waiting room
professional category | The day the patient waits in the imaging waiting room
Type of housing | The day the patient waits in the imaging waiting room
  house or building, floor, elevator, garden, ...
Lifestyle | The day the patient waits in the imaging waiting room
  urban, rural

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No